CLINICAL TRIAL: NCT03880864
Title: Application of Lung Ultrasound for Predicting Outcome of Weaning From Mechanical Ventilation
Brief Title: Lung Ultrasound for Predicting Outcome of Weaning From Mechanical Ventilation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Randa Ali Shoukry, Assistant Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FMASU R 12/2019
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Weaning Failure
Keywords: Lung ultrasound score; Weaning; Mechanical ventilation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Ultrasound — Lung ultrasound

SUMMARY:
Lung aeration loss can be measured via lung ultrasound, it is a non-invasive, bed side procedure, which can be performed rapidly and facilitates a dynamic assessment of lung aeration. Aim of the work: is to determine the role of lung ultrasound score as one of the predictors of successful weaning from mechanical ventilation in ICU patients.

DETAILED DESCRIPTION:
Patients should be assessed daily for their readiness to be weaned from mechanical ventilation, sedation must be withdrawn and all patients will be put on a spontaneous breathing trial (SBT), via T-piece, for 60 -120 minutes period, when they fulfil the weaning criteria. Patients who succeed to tolerate SBT will be extubated and monitored for signs of respiratory distress.

Clinical assessment during and after SBT:

* The ability of maintaining a respiration rate of less than 35/min, and keeping oxygen saturation more than 90%.
* Arterial blood gases (ABGs) will be done 30-60 minutes after SBT and after extubation.
* To detect signs of respiratory distress: diaphoresis, tachypnea (RR> 35/min), increase activity of accessory muscles of respiration, tachycardia (heart rate > 140 beats per minute), systolic blood pressure > 180 mmHg or <90 mmHg, appearance of new arrhythmia, or alteration in mental status (drowsiness or anxiety). ABGs: PaO2 ≤ 60 mmHg or oxygen saturation < 90% on FiO2 ≥ 0.4, PaCO2 > 50 mmHg, or an increase in by ≥ 8 mmHg, pH < 7.32 or a decrease in pH by ≥ 0.07 pH units.

Clinical assessment will be done by an intensivist who will be blinded to the LUS score results.

Lung ultrasound (LUS): will be performed while patients in supine position, with a curved probe on B- mode, using longitudinal view, to assess the amount of lung aeration. Each lung will be divided into anterior, lateral and posterior regions, each part will be divided to upper and lower zone, with total of 12 zones to undergo examination. Examination will be done by an expert physician in US.

Lung US score [9]: The 12 scanned regions will be summed to calculate the LUS score, which ranged from 0 and 36. In each zone, the worst ultrasound form will considered to be descriptive of the entire region.

* Score of 0: Normal aeration is signified by the presence of horizontal A lines, lung sliding, or less than 3 vertical B lines.
* Score of 1: moderate loss of aeration is characterized by multiple regularly or irregularly spaced B lines that originated from the pleural line.
* Score of 2: Severe loss of aeration is manifested by multiple coalescent B lines in several intercostal spaces of the specific zone. Detected in alveolar-interstitial syndrome.[
* Score of 3: Complete loss of aeration, as detected in lung consolidation or atelectasis, is characterized by tissue echogenicity, which is similar to liver or splenic tissues.

The score will be performed before starting and at the end of SBT (before extubation), or on developing respiratory distress during SBT.

Patients will be classified according to the possible outcome:

Successful weaning: patients who will not need re-intubation within 48 hours after extubation.

SBT failure: which will be diagnosed by the appearance of signs of respiratory distress during SBT and patients will be connected again to the ventilator. Extubation failure: will be defined as patients who developed signs of respiratory distress after extubation within 48hs and need reintubation or non-invasive ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* 50 adult patients over 18 years.
* Mechanically ventilated via an endotracheal tube for more than 24 hours.
* Patients that have an improvement in the underlying cause of respiratory failure.

Exclusion Criteria:

* Patients with tracheostomy
* Spinal cord injury above than T8
* Arrhythmias and or haemodynamic instability
* Patients having pneumothorax, or pneumomediastinum, chest tube or chest injuries.
* After thoracostomy, and pleural lesions or pleurodesis.
* Patients having severe chronic obstructive pulmonary disease (COPD) with forced expiratory volume less than 50% of predictive value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-12-02 (Estimated); Study Completion 2020-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with lung ultrasound score of less than 13 | 48 hours
  Successful weaning: patients who will not need re-intubation within 48 hours after extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Randa Ali Shoukry, Cairo, Al-Nozha, Egypt

IPD SHARING:
Plan to Share IPD: No